CLINICAL TRIAL: NCT00851136
Title: A Phase Ib Study of the Safety and Pharmacokinetics of PRO95780 Administered in Combination With the FOLFOX Regimen and Bevacizumab in Patients With Previously Untreated, Locally Advanced, Recurrent, and Metastatic Colorectal Cancer
Brief Title: A Study of PRO95780 Administered in Combination With the FOLFOX Regimen and Bevacizumab in Patients With Previously Untreated, Locally Advanced, Recurrent, and Metastatic Colorectal Cancer (APM4566g)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APM4566g
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: CRC; Colon cancer; Avastin; APM4566g
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Folfox protocol; drozitumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab; Drug: FOLFOX; Drug: PRO95780

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
Drug: FOLFOX — Intravenous repeating dose
Drug: PRO95780 — Intravenous repeating dose

SUMMARY:
This will be a multicenter, open-label study enrolling a total of up to 23 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CRC with evidence of locally advanced recurrent or metastatic disease and measurable tumor lesions
* Life expectancy > 3 months
* For patients of reproductive potential (males and females), use of reliable means for contraception throughout the trial and for 6 months following their final exposure to study treatment
* Willingness and capability to be accessible for study follow-up

Exclusion Criteria:

* Prior 5-FU, capecitabine, and/or oxaliplatin treatment with the exception of: prior oxaliplatin treatment≤ 6 weeks in the advanced or metastatic setting; prior treatment with 5-FU, capecitabine, and/or oxaliplatin in the adjuvant setting if relapse occurred > 6 months from concluding adjuvant therapy
* Peripheral neuropathy Grade ≥ 2
* Prior radiotherapy to a measurable metastatic lesion(s) to be used for response assessment, unless the lesion has progressed subsequent to the radiotherapy
* Radiotherapy to a peripheral lesion within 14 days prior to Cycle 1, Day 1, or radiotherapy to a thoracic, abdominal, or pelvic field within 28 days prior to Cycle 1, Day 1
* Chemotherapy, hormonal therapy, or immunotherapy within 4 weeks prior to Cycle 1, Day 1
* Evidence of clinically detectable ascites
* Other invasive malignancies within 5 years prior to Cycle 1, Day 1
* History or evidence upon physical examination of active central nervous system (CNS) disease
* Current or recent participation in another experimental drug study
* Clinically significant cardiovascular disease, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia within 1 year prior to Cycle 1, Day 1, or Grade II or greater peripheral vascular disease
* Active infection requiring parenteral antibiotics
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Cycle 1, Day 1, fine needle aspirations within 7 days prior to Cycle 1, Day 1, or anticipation of need for major surgical procedure during the course of the study
* Known or suspected to be positive for the human immunodeficiency virus (HIV)
* Known to be positive for hepatitis C or hepatitis B surface antigen
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of arterial thromboembolic event 6 months prior to Cycle 1, Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Cycle 1, Day 1
* Bleeding diathesis or coagulopathy
* Pregnancy (positive pregnancy test) or breast feeding
* Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities | Length and study

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events | Length of study
Change in vital signs | Length of study
Incidence and severity of infusion reactions | Length of study
Change in clinical laboratory results | Length of study
Incidence of anti-PRO95780 antibodies | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, M.D., Study Director — Genentech, Inc.